CLINICAL TRIAL: NCT02237573
Title: Impact of Handing to Patients With Viral Gastroenteritis or Upper Respiratory Tract Infections a Copy of the Consultation Report on Their Medicine Consumption: a Randomized Controlled Trial
Brief Title: Impact of Handing to Patients a Copy of the Consultation Report on Their Medicine Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Paris 7 - Denis Diderot (Other)
Responsible Party: Principal Investigator, TRAN Viet thi, assistant professor, University Paris 7 - Denis Diderot
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMG003
Record Dates: First submitted 2014-08-14; First posted 2014-09-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Viral Gastro Enteritis; Pharyngitis
Keywords: general practice; viral infections; consultation reports; drug prescription
MeSH Terms: conditions — Pharyngitis; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Written medical report and standardized medical advices
  Interventions: Other: Written medical report and standardized medical advices
- Control (Active Comparator): Standardized medical advice only
  Interventions: Other: Control

INTERVENTIONS:
Other: Written medical report and standardized medical advices — The intervention will include: 1) handing the patient at the end of the consultation a copy of the consultation report which will be composed of:
  1. a detailed report of the consultation (motive, case history, clinical examination, conclusion)
  2. written standardized medical advices from evidence published in the literature. Interventions will be designed by several general practitioners and tested by few patients.
  Arms: Intervention
Other: Control — Other:
  Oral standardized medical advices from evidence published in the literature. Physicians will be trained by a single investigator.
  Arms: Control

SUMMARY:
In France, patients with benign viral infections (ie: gastro enteritis and/or rhinopharyngitis, etc.) often receive several prescriptions from their doctors, although there is evidence that these medicines are not efficient.

We hypothesize that patients could be reassured by health advices, especially if they are written. In addition, we believe that doctors would feel less guilty for not prescribing drugs if they could hand written consultation reports to patients, in these situations.

We aim to assess the impact of handing to patients with viral gastroenteritis or upper respiratory tract infections, a copy of the consultation report on their medicine consumption.

DETAILED DESCRIPTION:
In France, 90% of General practitioners' (GPs) consultations end with prescription of drugs (versus only 43,2% in Netherlands). A french medical thesis published in 2013 showed that drugs prescriptions were not a priority for patients. Rather than medicine's prescription, patients preferred attentive listening associated with personalized advices from their GPs. Several studies also showed that a commercial relationship exists between doctors and patients. The prescription is like an exchange currency against the patient money.

We aim to assess the impact of handing to patients with viral gastroenteritis or upper respiratory tract infections, a copy of the consultation report on their medicine consumption.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with >18 ans Diagnosis of gastroenteritis or rhinopharyngitis by the physician Written consent by patient

Exclusion Criteria:

Patients who have already visited the doctor in the last 15 days A given patient can only be included once Diagnostic uncertainty or need of laboratory tests Cognitive impairment Only one patient by family or visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mean number of medications prescribed by the physician | 1 day
  We will assess the mean number of medications prescribed by the physician during the consultation.
  Two independent investigators will assess, aposteriori from medical records, each prescription to determine the number of prescribed drugs (including rhino pharyngeal desobstruction). In case of discrepancy in their assessments, a third investigator will help in consensus.

SECONDARY OUTCOMES:
Number (Proportion) of each class of prescribed drug | 1 day
  We will assess the frequency of each class of medications prescribed by the physician during the consultation.
  Classes will be: 1)paracetamol, 2)non steroidal anti inflammatory drug, 3)antibiotics, 4)physiological serum, 5)vasoconstrictor nasal spray, 6)oral spray, 7)cough syrup, 8)loperamide, 9)phloroglucinol, 10)antiemetic drugs, 11) antiseptic lozenges.
  Two independent investigators will assess each prescription made by physicians to determine the different prescribed drugs (including rhinopharyngeal desobstruction). In case of discrepancy in their assessments, a third investigator will help in consensus.
Number (Proportion) of reconsultation | 30 days
  A single investigator will recontact all included patients by telephone to assess if they reconsulted a doctor for the same motive in the period. If they cannot be contacted by phone, they will be contacted by e-mail. A second call will be done after 7 days in case they did not answer the first call.
  We will compare proportion of reconsultation between the two groups.
Number (Proportion) of patients resorting to self-treatment | 30 days
  A single investigator will recontact all included patients by telephone to assess if included patients self treated themselves using drugs they had at their disposal or using non prescription drugs. If they cannot be contacted by phone, they will be contacted by e-mail. A second call will be done after 7 days in case they did not answer the first call.
  We will compare proportion of self treatment between the two groups
Number (Proportion) of adverse effects | 30 days
  One investigator will assess, aposteriori from medical records, if patients reconsulted for a motive that could be associated with an aggravation of the viral infection (gastro enteritis or rhinopharyngitis).
  In addition, all included patients will be recontacted by telephone (or e-mail in case they do not answer the phone) We will assess nature and number of cases.

CONTACTS AND LOCATIONS:
Overall Officials: Viet-Thi Tran, MD, Principal Investigator — Paris Diderot University
Locations (1):
- Faculté Xavier Bichat, Paris, France

REFERENCES:
- [Background] Macfarlane J, Holmes W, Gard P, Thornhill D, Macfarlane R, Hubbard R. Reducing antibiotic use for acute bronchitis in primary care: blinded, randomised controlled trial of patient information leaflet. BMJ. 2002 Jan 12;324(7329):91-4. doi: 10.1136/bmj.324.7329.91. PMID 11786454